CLINICAL TRIAL: NCT06894030
Title: Investigating the Longitudinal Efficacy of Cognitive Cueing and Video Intervention for Gait in People With Parkinson's Disease
Brief Title: Cognitive Cueing and Video Intervention for Gait in Parkinson's Disease
Acronym: CogCueVidPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Jeffrey Holmes, Associate Professor, School of Occupational Therapy, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HSREB125635
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease
Keywords: Gait; Cueing; Balance; Mobility
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The Video Start group will receive their gait training video once the intervention begins. The Video Delay group will receive their gait training video after a 4-week delay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video Start (Experimental)
  Interventions: Behavioral: Gait Training Video; Behavioral: Cognitive Cue
- Video Delay (Experimental)
  Interventions: Behavioral: Gait Training Video; Behavioral: Cognitive Cue

INTERVENTIONS:
Behavioral: Gait Training Video — Personalized gait training videos featuring cued and non-cued gait for participants
Behavioral: Cognitive Cue — A verbal cue to be mentally rehearsed by each participant

SUMMARY:
The goal of this clinical trial is to learn if cognitive cueing (eg., prompting individuals to think about taking big-long steps while walking), either as a stand- alone intervention or combined with a personalized gait training video, can improve gait (walking), mobility, and balance confidence for individuals with Parkinson's Disease. The main questions it aims to answer are:

1. Does focusing on cognitive cues while walking improve gait, mobility, and balance confidence for individuals with Parkinson's Disease?
2. Does incorporating a personalized gait training video alongside cognitive cueing lead to amplified improvements in gait, mobility, and balance confidence for individuals with Parkinson's Disease?

Researchers will compare how gait, mobility, balance confidence and quality of life change over time for participants when they practice walking with and without a cognitive cue alone, and when they practice with using a personalized gait training video.

The researchers are also interested in how participation in this trial will affect quality of life and conscious attention to gait.

Participants will

* Complete walking trials on an instrumented mat that records data on their walking ability. These trials will be undertaken without a cognitive cue and while participants mentally rehearse a series of 3 cognitive cues (Take big long steps; Walk heel-toe; Stand up straight).
* Be informed about which of the 3 cues best improved their walking and will receive a personalized gait training video for at home practice.
* Complete online surveys that ask questions about their Parkinson's Disease, mobility, balance confidence quality of life and conscious attention to gait.
* Visit the research facility 3 to 4 times during the study to have their gait (walking), mobility, balance confidence, quality of life and conscious attention to gait assessed and reassessed.
* Practice both with and without their personalized video at home and keep a diary to record their practice sessions
* Participate in a brief interview to discuss their experiences with the training and their perceptions of the effectiveness of cognitive cues and video-recorded feedback

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with Parkinson's Disease
* Be fluent in English
* Be able to walk independently and without a walking aid for at least 10 minutes
* Have no other cognitive or neurological impairments (e.g., brain tumours, recent concussion, stroke, brain injury)

Exclusion Criteria:

* Deep Brain Stimulation (DBS) implant
* Standardized Mini Mental State Examination (SMMSE) score less than 24

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Mean Stride Length | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Mean of stride length measured in centimeters (cm).
Variability iin Stride Length | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Coefficient of variation in stride length.
Mean of Stride Width | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Mean of stride width measured in centimeters (cm).
Variability in Stride Width | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Coefficient of variation in stride width.
Mean of Stride Velocity | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Mean of stride velocity measured in centimeters per second-squared (cm/s^2).
Variability in Sride Velocity | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Coefficient of variation in stride velocity.
Mean of Double Support Time | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Mean double support time measured as a proportion (0-1). This is the proportion of a gait cycle spent with two feet on the ground.
Variability in Double Support Time | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Coefficient of variation in double support time
Timed Up and Go (TUG) | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  Timed test of functional mobility where participants are recorded on the number of seconds it takes to stand up from a chair, walk 10ft, turn around, walk back 10ft, and sit back in the chair. Longer times suggest lower functional mobility.

SECONDARY OUTCOMES:
Activities-specific Balance Confidence Scale (ABC) | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  16-item self-report scale where participants rate their confidence on items using 0 to 100 scale. The scale score is the mean of all items, with a maximum of 100 and minimum of 0. Higher score indicate greater balance confidence.
Gait-Specific Attentional Profile (G-SAP) | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  11-item self-report scale where participants rate the frequency that they experience the scenarios described by the items on a 5pt Likert scale (0- not all all, 5 - very much so). Scores are calculated on the followings 4 sub-scales ( Anxiety [/15], Conscious movement processing[/15], Fall-related ruminations[/10], Processing efficiency[/10]). Lower sum scores for Anxiety, Fall related ruminations and Processing efficiency indicate better outcomes. Higher sum score for Conscious movement processing indicate greater attention is focused on walking.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | From baseline to the end of the study (~17 weeks after baseline) as follows: Week 0 (Baseline), Week 5 (Session 2); Week 9 (Session 3 Video Delay Group ONLY); Week 13 (Session 3 Video Start Group ONLY); Week 17 (Session 4 Video Delay Group ONLY)
  39-item self-report scale designed to evaluate quality of life of people with Parkinson's Disease across 8 dimensions of daily living. Participants rank items on a 5pt Likert scale (0 - never, 4 - always). Higher scores in each dimension's sub-scale and the scale as a whole indicate a poorer quality of life.
Standardized Mini Mental State Examination (SMMSE) | At baseline only
  11 items/tasks administered to measure participant's cognitive abilities and screen for potential cognitive impairment. The final score is out of 30 total pts where higher scores indicate greater cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Brain and Mind, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided